CLINICAL TRIAL: NCT02510222
Title: Effect of Magnesium Therapy on Spasticity and Constipation in Children With Cerebral Palsy
Brief Title: Magnesium Therapy in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sahar M.A. Hassanein, MD, Professor of Pediatrics , Faculty of Medicine, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pediatrics MS
Record Dates: First submitted 2015-07-26; First posted 2015-07-29 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Cerebral Palsy
Keywords: child
MeSH Terms: conditions — Cerebral Palsy | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Magnesium sulfate (Experimental): Magnesium sulphate 4% concentration orally ( 65 mg per day for children one to three years of age; 110 mg per day for children four to eight years of age; 350 mg per day for children older than eight years) for 1 month
  Interventions: Dietary Supplement: Oral magnesium sulfate
- Control (Placebo Comparator): Fifty children with cerebral palsy will be treated with conventional therapy as physiotherapy. They will receive placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Oral magnesium sulfate — Magnesium sulfate 4% concentration in a dose of 65 mg/day for infants and children aged 1-3 years , 110 mg/day for those 3-8 years and 350 mg/day for those above 9 years .Each 1 ml of the magnesium sulfate used contains 0.325 mEq (milliequivalent) of elemental magnesium which equals to 4 mg elemental magnesium .
  Arms: Oral Magnesium sulfate
Other: Placebo
  Arms: Control

SUMMARY:
This study is considered a pilot exploratory study. Intervention, prospective, double-armed, randomized, placebo-control clinical trial.

The therapeutic effect of oral Magnesium sulfate on spasticity and constipation will be studied.

DETAILED DESCRIPTION:
Spasticity and constipation are major problems hindering improvement in motor development in children with cerebral palsy.

Decreasing spasticity will have a positive effect on motor development and quality of life for the child and his family.

The aim is to study the therapeutic and adverse effects of oral magnesium sulfate therapy on spasticity and constipation in infants and children with cerebral palsy.

Hundred children with spastic cerebral palsy will be randomized to either intervention group n=50 will be treated with magnesium sulfate 4% orally for 28 days to treat spasticity and constipation in addition to their conventional treatment, or placebo group n=50 will receive conventional treatment and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age below12 years.
* Presence of spasticity without joint contracture Spasticity is defined as velocity dependent, increased resistance to passive muscle stretch.
* Acceptance of caregivers to participate in the study and signing the written consent.
* Constipation will be defined according to Rome lll criteria.presence of at least 2 of the following 2 motions week, history of painful or hard bowel movement, presence of large diameter stools that stools that may obstruct the toilets (Burgers et al., 2012).

Exclusion Criteria:

* Severe growth retardation (Below the 10th centile for weight and length charts children with cerebral palsy).
* Gastrostomy tube feeding.
* Joint contractures.
* Congenital malformations.
* Suspected inborn error of metabolism.
* Suspected inherited neurologic disease.
* Care giver's refusal to participate in the study.
* Occurrence of side effects of oral magnesium sulfate.
* Patients with cardiac, renal, GIT problem or chronic diarrhea.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Decrease in muscle tone evaluated by Modified Ashworth Index and constipation ROM-lll criteria | 1 month

SECONDARY OUTCOMES:
Improvement in H/M ratio in H-reflex by electrophysiologic assessment | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Sahar MA Hassanein, PhD, MD, Principal Investigator — Pediatric department, Faculty of Medicine , Ain Shams University
Locations (1):
- Children's Hospital, Faculty of Medicine, Ain Shams University, Cairo, Cairo Governorate, Egypt